CLINICAL TRIAL: NCT06116435
Title: Designing With Dissemination in Mind: Development and Evaluation of a Theory-based Physical Activity Intervention Using the Multiphase Optimization Strategy: Aim 2
Brief Title: A Pilot Factorial Trial of an Integrated Lifestyle Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 23-1154; K01HL161417 (NIH)
Record Dates: First submitted 2023-10-12; First posted 2023-11-03 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Physical Inactivity; Overweight and Obesity
Keywords: physical activity; obesity; weight loss; nutrition; diet; lifestyle intervention
MeSH Terms: conditions — Sedentary Behavior; Overweight; Obesity; Motor Activity; Weight Loss | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: 2x2x2 full factorial pilot randomized trial
Who Masked: Outcomes Assessor
Masking Description: Trials participants will know their intervention condition as will the lay coach involved in delivering the intervention. Assessors measuring body composition (DXA), self-reported energy intake, and metabolic parameters will be blinded to participant condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- PreventT2 + Move group-based classes (Experimental): Participants will receive a 6-month lifestyle weight management program based on the publicly available Prevent T2 curriculum (formally known as the National Diabetes Prevention Program), integrated with the Move group-based classes. Group classes will be delivered weekly in weeks 1-12, and biweekly in weeks 13-26. Group-based classes will be taught virtually by a trained Registered Dietitian from the Colorado Nutrition Obesity Research Center Clinical Intervention and Translation (CIT) Core.
  Interventions: Behavioral: Prevent T2; Behavioral: Move group-based classes
- PreventT2 + Move group-based classes + Fitness Membership (Experimental): Participants will receive a 6-month lifestyle weight management program based on the publicly available Prevent T2 curriculum (formally known as the National Diabetes Prevention Program), integrated with the Move group-based classes. Group classes will be delivered weekly in weeks 1-12, and biweekly in weeks 13-26. Group-based classes will be taught virtually by a trained Registered Dietitian from the Colorado Nutrition Obesity Research Center Clinical Intervention and Translation (CIT) Core. Participants will also receive a 6-month membership to the Peloton fitness app.
  Interventions: Behavioral: Prevent T2; Behavioral: Move group-based classes; Behavioral: Fitness Membership
- PreventT2 + Move group-based classes + Mental Imagery (Experimental): Participants will receive a 6-month lifestyle weight management program based on the publicly available Prevent T2 curriculum (formally known as the National Diabetes Prevention Program), integrated with the Move group-based classes. Group classes will be delivered weekly in weeks 1-12, and biweekly in weeks 13-26. Group-based classes will be taught virtually by a trained Registered Dietitian from the Colorado Nutrition Obesity Research Center Clinical Intervention and Translation (CIT) Core. In addition, participants will receive access to online mental guided imagery sessions. Guided positive exercise imagery scripts were developed based on work from Williams et al. and prompt several sensory and emotional experiences.
  Interventions: Behavioral: Prevent T2; Behavioral: Move group-based classes; Behavioral: Mental Imagery
- PreventT2 + Move group-based classes + Mental Imagery + Fitness Membership (Experimental): Participants will receive a 6-month lifestyle weight management program based on the publicly available Prevent T2 curriculum (formally known as the National Diabetes Prevention Program), integrated with the Move group-based classes. Group classes will be delivered weekly in weeks 1-12, and biweekly in weeks 13-26. Group-based classes will be taught virtually by a trained Registered Dietitian from the Colorado Nutrition Obesity Research Center Clinical Intervention and Translation (CIT) Core. Participants will also receive a 6-month membership to the Peloton fitness app. In addition, participants will receive access to online mental guided imagery sessions. Guided positive exercise imagery scripts were developed based on work from Williams et al. and prompt several sensory and emotional experiences.
  Interventions: Behavioral: Prevent T2; Behavioral: Move group-based classes; Behavioral: Fitness Membership; Behavioral: Mental Imagery
- PreventT2 + Move group-based classes + Move 1:1 Support (Experimental): Participants will receive a 6-month lifestyle weight management program based on the publicly available Prevent T2 curriculum (formally known as the National Diabetes Prevention Program), integrated with the Move group-based classes. Group classes will be delivered weekly in weeks 1-12, and biweekly in weeks 13-26. Group-based classes will be taught virtually by a trained Registered Dietitian from the Colorado Nutrition Obesity Research Center Clinical Intervention and Translation (CIT) Core. Participants will also receive Move individualized support sessions. The 1:1 support sessions are designed to help participants adopt the physical activity messages from each Move group-based class into their daily lives.
  Interventions: Behavioral: Prevent T2; Behavioral: Move group-based classes; Behavioral: Move 1:1 Support
- PreventT2 + Move group-based classes + Fitness Membership + Move 1:1 Support (Experimental): Participants will receive a 6-month lifestyle weight management program based on the publicly available Prevent T2 curriculum (formally known as the National Diabetes Prevention Program), integrated with the Move group-based classes. Group classes will be delivered weekly in weeks 1-12, and biweekly in weeks 13-26. Group-based classes will be taught virtually by a trained Registered Dietitian from the Colorado Nutrition Obesity Research Center Clinical Intervention and Translation (CIT) Core. Participants will also receive a 6-month membership to the Peloton fitness app. Participants will also receive Move individualized support sessions. The 1:1 support sessions are designed to help participants adopt the physical activity messages from each Move group-based class into their daily lives.
  Interventions: Behavioral: Prevent T2; Behavioral: Move group-based classes; Behavioral: Fitness Membership; Behavioral: Move 1:1 Support
- PreventT2 + Move group-based classes + Mental Imagery + Move 1:1 Support (Experimental): Participants will receive a 6-month lifestyle weight management program based on the publicly available Prevent T2 curriculum (formally known as the National Diabetes Prevention Program), integrated with the Move group-based classes. Group classes will be delivered weekly in weeks 1-12, and biweekly in weeks 13-26. Group-based classes will be taught virtually by a trained Registered Dietitian from the Colorado Nutrition Obesity Research Center Clinical Intervention and Translation (CIT) Core. Participants will also receive Move individualized support sessions. The 1:1 support sessions are designed to help participants adopt the physical activity messages from each Move group-based class into their daily lives. In addition, participants will receive access to online mental guided imagery sessions. Guided positive exercise imagery scripts were developed based on work from Williams et al. and prompt several sensory and emotional experiences.
  Interventions: Behavioral: Prevent T2; Behavioral: Move group-based classes; Behavioral: Mental Imagery; Behavioral: Move 1:1 Support
- PreventT2 + Move group-based classes + Fitness Membership + Mental Imagery + Move 1:1 Support (Experimental): Participants will receive a 6-month lifestyle weight management program based on the publicly available Prevent T2 curriculum, integrated with the Move group-based classes. Group classes will be delivered weekly in weeks 1-12, and biweekly in weeks 13-26. Group-based classes will be taught virtually by a trained Registered Dietitian. Participants will also receive a 6-month membership to the Peloton fitness app. Participants will also receive Move individualized support sessions. In addition, participants will receive access to online mental guided imagery sessions.
  Interventions: Behavioral: Prevent T2; Behavioral: Move group-based classes; Behavioral: Fitness Membership; Behavioral: Mental Imagery; Behavioral: Move 1:1 Support

INTERVENTIONS:
Behavioral: Prevent T2 — The PreventT2 curriculum is based on the original 2002 Diabetes Prevention Prevention (DPP) trial and follow-up studies. It promotes modest weight loss (5-7%) and increased physical activity through a lifestyle change program and also reflects new literature on self-efficacy, physical activity, and diet. There are 16 modules that will be delivered over 6 months. Participants will receive a calorie goal and be asked to count calories in order to reduce their caloric intake.
Behavioral: Move group-based classes — The Move physical activity support program group-based classes are based on Self-Determination Theory and encourage improvements in autonomous motivation for physical activity. These group-based classes are integrated within the Prevent T2 program curricula.
Behavioral: Fitness Membership — Participants will receive 6 months of the Peloton fitness membership. This includes access to livestream and on-demand fitness classes including walking, strength training, yoga, meditation, stretching, etc.
  Arms: PreventT2 + Move group-based classes + Fitness Membership; PreventT2 + Move group-based classes + Fitness Membership + Mental Imagery + Move 1:1 Support; PreventT2 + Move group-based classes + Fitness Membership + Move 1:1 Support; PreventT2 + Move group-based classes + Mental Imagery + Fitness Membership
Behavioral: Mental Imagery — Participants will receive access to positive mental guided imagery recordings. Recordings describe a pleasant experience while walking and range from 2-8 minutes in duration.
  Arms: PreventT2 + Move group-based classes + Fitness Membership + Mental Imagery + Move 1:1 Support; PreventT2 + Move group-based classes + Mental Imagery; PreventT2 + Move group-based classes + Mental Imagery + Fitness Membership; PreventT2 + Move group-based classes + Mental Imagery + Move 1:1 Support
Behavioral: Move 1:1 Support — Participants will meet individually with their class instructor to receive personalized recommendations on how to incorporate messages from the Move group-based classes into their daily lives. Sessions are based on Self-Determination Theory and will last approximately 45 minutes.
  Arms: PreventT2 + Move group-based classes + Fitness Membership + Mental Imagery + Move 1:1 Support; PreventT2 + Move group-based classes + Fitness Membership + Move 1:1 Support; PreventT2 + Move group-based classes + Mental Imagery + Move 1:1 Support; PreventT2 + Move group-based classes + Move 1:1 Support

SUMMARY:
This study plans to learn more about the feasibility and acceptability of integrating the Move physical activity support program within an existing lifestyle intervention program.

ELIGIBILITY:
Inclusion Criteria:

* For all types of research participants:

  * Men and Women
  * Age 18-65 years
  * Have access to a computer and/or smart phone, and Wi-Fi
  * Speak English (since all study materials are in English and the intervention will be delivered in a group-class setting with a coach who speaks English, we are only able to accommodate English-speakers at this time)
* For the patient participants only:

  * Body Mass Index 25-45 kg/m2
  * Insufficiently active (defined as <150 min/week of voluntary exercise at moderate intensity over the past 3 months)
  * Willing not to enroll in any other formal weight loss, or physical activity program over the next 5 months.
  * Have a primary care physician (or has access to a healthcare professional and/or are willing to establish care with a primary care physician prior to study enrollment) to address medical issues which may arise during screening or study procedures/interventions.
  * Capable and willing to give informed consent, understand exclusion criteria, attend the Move program sessions, and complete outcome measures.
* For the provider participants only:

  * >1 year experience with delivering lifestyle interventions involving changes in diet and/or exercise behaviors.

Exclusion Criteria:

* For patient participants:

  * Considered high risk, based on the American College of Sports Medicine Guidelines for Exercise Testing and Prescription (i.e. have cardiovascular disease symptoms or known cardiovascular disease, diabetes, or end-stage renal disease).
  * Females who are currently pregnant or lactating, were pregnant within the past 3 months, or planning to become pregnant in the next 5 months will also be excluded
  * Self-reported cardiovascular disease:
  * Cardiac, peripheral vascular, or cerebrovascular disease
  * Self-reported symptoms suggestive of cardiovascular disease: pain, discomfort in the chest, neck, jaw, arms, or other areas that may result from cardiac ischemia; shortness of breath at rest or with mild exertion; dizziness or syncope; orthopnea or paroxysmal nocturnal dyspnea; ankle edema; palpitations or tachycardia; intermittent claudication
  * Self-reported end-stage renal disease
  * Self-reported diabetes (history of type 1 or type 2 diabetes)
  * Uncontrolled hypertension, defined as diastolic blood pressure >100 mmHG, systolic blood pressure >160 mmHG, or resting heart rate >100 bpm as measured in duplicate at the screening visit after 5 minutes of rest in a seated position.
  * Self-reported pulmonary disease requiring chronic oxygen supplementation; severe asthma or chronic obstructive pulmonary disease requiring hospitalization in past year.
  * Plans to relocate in the next 16 months
  * Currently participating in or planning to participate in any formal weight loss, dietary modification, or physical activity/exercise programs or clinical trials.
  * Current severe depression or history of severe depression within the previous year, based on Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria for Major Depressive Episode. Score > 18 on Beck Depression Inventory (BDI) will require further assessment by the Study Medical Doctor (MD) to determine if it is appropriate for the subject to participate in the study.
  * History of other significant psychiatric illnesses (e.g., psychosis, schizophrenia, mania, bipolar disorder) which in the opinion of the Study MD would interfere with ability to adhere to the exercise intervention.
  * History of clinically diagnosed eating disorders including anorexia nervosa, bulimia, binge eating disorder. Score >20 on the Eating Attitudes Test (EATS-26) or pattern of response on the Questionnaire on Eating and Weight Patterns-5 (QEWP-5) suggestive of possible binge eating disorder or bulimia will require further assessment by the Study MD to determine if it is appropriate for the subject to participate in the study.
  * Current alcohol or substance abuse
  * Nicotine use (current or past 6 months)
  * Regular use of prescription or over-the-counter medications known to significantly impact appetite, weight, sleep, or energy metabolism (e.g., appetite suppressants, lithium, stimulants, anti-psychotics, tricyclic antidepressants)
  * Regular use of obesity pharmacotherapeutic agents within the last 6 months.
  * Previous obesity treatment with surgery or weight loss device, except: (1) liposuction and/or abdominoplasty if performed > 1 year before screening, (2) lap banding if the band has been removed > 1 year before screening, (3) intragastric balloon if the balloon has been removed > 1 year before screening (4) duodenal-jejunal bypass sleeve, if the sleeve has been removed > 1 year before screening or 5) AspireAssist or other endoscopically placed weight loss device if the device has been removed > 1 year before screening.
  * Currently has access to and uses a fitness membership (defined as having used membership within the past month)
* For provider participants:

  * None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the Move physical activity support program - Qualitative | 6 months
  Acceptability of the Move physical activity support program will be assessed with results of the semi-structured focus groups or interviews from the participant and provider perspectives.
Feasibility of the Move physical activity support program - Qualitative | 6 months
  Feasibility of the Move physical activity support program will be assessed with results of the semi-structured focus groups or interviews from the participant and provider perspectives.

SECONDARY OUTCOMES:
Acceptability of the Move physical activity support program components - Quantitative | 6 months
  Acceptability of the integrated Move physical activity support program components will be assessed using the Net Promoter Score (NPS) from the participant and provider perspectives. Scores range from -100 to +100, with higher scores indicating a better outcome.
Feasibility of the Move physical activity support program - Quantitative | 6 months
  Feasibility of the Move physical activity support program will be assessed using the Perceived Characteristics of Intervention Scale (PCIS) collected only at the level of the provider. Scores range from 0 to 4, with higher scores indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Ostendorf, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No